CLINICAL TRIAL: NCT04210765
Title: The Effect of Incremental Clomiphene Citrate(CC) Doses in Successive Induction Cycles on the Endogenous Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH) and Steroid Hormone Responses to Treatment
Brief Title: Incremental Clomiphene Citrate Doses in Successive Cycles and FSH, LH and Steroid Hormone Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019.08.1.04.061
Record Dates: First submitted 2019-12-13; First posted 2019-12-26 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2019-12

CONDITIONS: Unexplained Infertility; Ovulation Disorder
Keywords: infertility; unexplained infertility; ovulation induction; clomiphene citrate
MeSH Terms: conditions — Infertility | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clomiphene citrate group 1 (Active Comparator): Clomiphene citrate dose 50mg/day for 5 days starting on cycle day (2-4).
  Interventions: Drug: Clomiphene Citrate
- Clomiphene citrate group 2 (Active Comparator): Non-responsive to ovulation induction with Clomiphene Citrate with dose:50mg/day; and treated with dose:100mg/day in the succeeding cycle for 5 days, starting on cycle day (2-4).
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Clomiphene Citrate — Clomiphene citrate used in incremental doses in nonresponsive cases.
  Other Names: CC

SUMMARY:
This study was planned to assess the initial and endogenous FSH, LH and steroid responses to incremental CC doses in successive ovulation induction cycles to treat anovulation in patients with unexplained infertility.

DETAILED DESCRIPTION:
In the Bagcilar Research and Training Hospital Obstetrics and Gynecology department outpatient clinic for infertility, the basal gonadotropin and androgen levels are routinely measured. In unexplained infertility couples with normal ovarian reserves the first line drug used for ovulation induction is CC. The starting dose is 50mg/day and the treatment is started within the 2nd to the 5th days of the menstrual cycle and continued for 5 days. Starting on the 2nd-3rd day following the last dose of the drug, the follicular growth was monitored with the transvaginal ultrasound and blood levels of hormones including FSH, LH, estradiol, progesterone, androstenedione, testosterone, and dehydroepiandrosterone sulphate were measured every 2-3 days. In this follow-up, if no follicular growth was observed day21 of the cycle, the CC dose was increased to CC 100mg/day (2X1, 50mg). If follicular growth and ovulation is achieved with no concluding conception, the same dose of CC is used in the following 2-3 cycles. When a maximum number of 2 dominant follicles are obtained ovulation is triggered with recombinant human chorionic gonadotropin (rhCG) and timed coit or intrauterine insemination is conducted.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years of age
* unexplained infertility
* first-line treatment
* Normal or increased ovarian reserve
* lack of ovulatory response to CC 50mg for 5 days

Exclusion Criteria:

* Male factor
* Tubal Factor
* Severe endometriosis
* Previous ovarian surgery

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with unexplained infertility
Enrollment: 50 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Changes in the endogenous blood levels of FSH, LH in successive cycles | Menstrual cycle at day 3 and day 9 and the trigger day respectively (each cycle is 28 days
  FSH (mIU/ml), LH (mIU/ml) blood levels measured with Enzyme-Linked ImmunoSorbent Assay (ELISA) tests.
Changes in the endogenous blood levels of steroids (including Androstenedione, Progesterone, Testosterone, estradiol) in successive cycles | Menstrual cycle at day 3 and day 9 and the trigger day respectively (each cycle is 28 days)
  Blood levels of steroids: Androstenedione (ng/ml), Progesterone (ng/ml), Testosterone (ng/ml), estradiol (pg/ml) measured with ELISA tests.

SECONDARY OUTCOMES:
conception rate | 15-20 days following intrauterine insemination.
  beta-hCG (IU/L)measured with ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim E Kovalak, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Teaching and Research Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozyurek ES, Yoldemir T, Artar G. Androstenedione response to recombinant human FSH is the most valid predictor of the number of selected follicles in polycystic ovarian syndrome: (a case-control study). J Ovarian Res. 2017 May 12;10(1):34. doi: 10.1186/s13048-017-0330-7. PMID 28494798
- [Background] Hager M, Horath S, Frigo P, Koch M, Marculescu R, Ott J. Changes in serum markers of patients with PCOS during consecutive clomiphene stimulation cycles: a retrospective study. J Ovarian Res. 2019 Oct 4;12(1):91. doi: 10.1186/s13048-019-0564-7. PMID 31585548